CLINICAL TRIAL: NCT01066910
Title: Parents As The Agent Of Change For Childhood Obesity (PAAC)
Acronym: PAAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0611M96906
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Obesity
Keywords: Obesity; Childhood Obesity; Exercise; Nutrition
MeSH Terms: conditions — Obesity; Pediatric Obesity; Motor Activity | interventions — Behavior Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Parent-only (Experimental)
  Interventions: Behavioral: Behavioral treatment for childhood obesity
- Parent and child (Active Comparator)
  Interventions: Behavioral: Behavioral treatment for childhood obesity

INTERVENTIONS:
Behavioral: Behavioral treatment for childhood obesity — Behavioral treatment for childhood obesity includes nutrition and physical activity recommendations, and behavior therapy skills for parent and child.
  Arms: Parent-only
Behavioral: Behavioral treatment for childhood obesity — Behavioral treatment for childhood obesity includes nutrition and physical activity recommendations, and behavior therapy skills for parent and child.
  Arms: Parent and child

SUMMARY:
The objective of this study is to test and evaluate the effectiveness of a parent-only treatment for childhood obesity. This study provides state-of-the-art treatment for childhood obesity. Parents and children will participate in treatment groups for 6 months. These treatment groups include recommendations to decrease overall caloric intake (by increasing fruits and vegetables), increasing physical activity, decreasing sedentary behavior and changing the home food environment. We are currently implementing this treatment in the Healthy Choices Program which is part of the Childhood Obesity Clinic at the University of Minnesota. Len Epstein at the University of Buffalo has been publishing on this treatment protocol for 30 years.

DETAILED DESCRIPTION:
The objective of this study is to pilot test and evaluate the efficacy of a parent-only treatment for childhood obesity. The central working hypothesis is that the parent-only treatment will result in greater weight loss for the overweight child as compared to the parent + child treatment. The specific aims of this application focus on comparing a behavioral parent-only intervention to a parent + child intervention for childhood obesity.

The primary aim of the proposed study is to compare the efficacy of the parent-only treatment to the parent + child treatment for childhood obesity.

The secondary aim is to compare treatment groups on change in the child and parent diet and exercise behavior, change in the home food environment, and parent weight post-treatment and at 6-months post-treatment.

This study is a randomized, clinical pilot trial evaluating two 6-month treatments for childhood obesity; parent + child and parent-only groups, with 6-months of post-treatment follow-up. The two treatments will differ in terms of the designated recipient of treatment, which will be delivered either to parents-only or to parents and children separately. Study outcomes will be assessed at baseline, immediately post-treatment, and 6-months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* An overweight child (>95th%) in the family who is between the ages of 8-12.
* A parent willing to participate and attend all treatment meetings.
* Family willing to commit to 6 months of treatment attendance, and follow-up for 6 months post-treatment.
* Family willing to submit the $60 deposit.

Exclusion Criteria:

* Child psychiatric disorder diagnoses (based on parent report).
* Child diagnoses of a serious current physical disease (such as diabetes) for which physician supervision of diet and exercise prescription are needed.
* Family with restrictions on types of food, such as food allergies, or religious or ethnic practices that limit the foods available in the home.
* Child with physical difficulties that limit the ability to exercise.
* Child with an active eating disorder.

All exclusionary and inclusionary criteria are similar to those in previous studies of Epstein and colleagues and Golan and colleagues.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2006-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Child BMI percentile, Child BMI, Child BMI_Z | 11 months

SECONDARY OUTCOMES:
Parent BMI, Child nutritional intake, Child physical activity | 11 months

CONTACTS AND LOCATIONS:
Overall Officials: Kerri N Boutelle, Ph.D., L.P., Principal Investigator — University of Minnesota - Dept of Pediatrics
Locations (1):
- KDWB University Pediatrics Family Center (UMP Stand alone clinic), Minneapolis, Minnesota, United States